CLINICAL TRIAL: NCT05477641
Title: Analgesic Comparison of Pericapsular Nerve Group (PENG) Block and Lateral Femoral Cutaneous Nerve (LFCN) Block to Fascia Iliaca Compartment Block (FICB) in Patients Undergoing Primary Total Hip Arthroplasty (THA).
Brief Title: Analgesic Comparison of PENG/LFCN to FICB for Total Hip Arthroplasty
Acronym: PengvsFICB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SSM Health Bone and Joint Hospital at St Anthony (Other)
Responsible Party: Principal Investigator, Patrick Myer, Chief CRNA SSM Bone and Joint Hospital, SSM Health Bone and Joint Hospital at St Anthony
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00060032
Record Dates: First submitted 2022-01-27; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, controlled study
Who Masked: Participant
Masking Description: Patient will be randomized into one of the 2 groups, but will not know which group. Also, the insertion site for both techniques is similar, so they won't be able to tell which group form that evidence either.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pericapsular nerve group block and lateral femoral cutaneous nerve block (Active Comparator): Nerve blocks
  Interventions: Procedure: Pericapsular Nerve Group Block with Lateral Femoral Cutaneous Nerve Block; Procedure: Fascia Iliaca Compartment Block
- fascia iliaca compartment block (Active Comparator): Nerve block
  Interventions: Procedure: Pericapsular Nerve Group Block with Lateral Femoral Cutaneous Nerve Block; Procedure: Fascia Iliaca Compartment Block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block with Lateral Femoral Cutaneous Nerve Block — Local anesthetic will be deposited along the lower pelvis to block 3 nerves that innervate the anterior hip capsule
Procedure: Fascia Iliaca Compartment Block — Local anesthetic is deposited between the fascia iliaca and the internal oblique muscle in an attempt to block 3 nerves that innervate the hip.
  Other Names: Suprainguinal Fascia Iliaca Block

SUMMARY:
This study compares 2 commonly used interventions (regional pain blocks) used in hip arthroplasty for pain control. One of the interventions is newer and not widely established.

DETAILED DESCRIPTION:
This study will compare the FICB to the PENG/LFCN blocks. Patient reported pain scores on a verbal numeric rating scale will be utilized and recorded in the PACU and postoperatively at 3, 6, 12, 18, 24, 36 and 48 hours after patient arrival in the PACU. Additionally, opioid consumption will be converted to morphine milliequivalents and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria for the study were: age 40-80, Physical Status I-III, BMI less than 40 kg/m2, ability to read and speak English, able to sign their own consent form and undergoing elective primary total hip arthroplasty.

Exclusion Criteria:

* Patients were excluded if they were chronically prescribed opioids for a condition unrelated to their surgical hip pain, were deemed Physical Status 4 or higher, had an ongoing coagulopathy, had any infection near the site of injection, had an allergy to local anesthetics, deemed to have diabetic neuropathy, deemed to have a contraindication to spinal anesthesia or were unable to report their pain scores reliably (as in severe dementia or similar).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Verbal Numeric Pain Score Comparison of Pericapsular Nerve Group (PENG) Block and Lateral Femoral Cutaneous Nerve (LFCN) Block to Fascia Iliaca Compartment Block (FICB) in Patients Undergoing Primary Total Hip Arthroplasty (THA). | 1 year
  Patient reported pain scores will be monitored and tracked and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- SSM Healthcare Bone and Joint Hosptial at St Anthony, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedard NA, Elkins JM, Brown TS. Effect of COVID-19 on Hip and Knee Arthroplasty Surgical Volume in the United States. J Arthroplasty. 2020 Jul;35(7S):S45-S48. doi: 10.1016/j.arth.2020.04.060. Epub 2020 Apr 24. PMID 32381441
- [Background] Berlioz BE, Bojaxhi E. PENG Regional Block(Archived). 2024 Oct 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK565870/ PMID 33351429
- [Background] Soffin EM, YaDeau JT. Enhanced recovery after surgery for primary hip and knee arthroplasty: a review of the evidence. Br J Anaesth. 2016 Dec;117(suppl 3):iii62-iii72. doi: 10.1093/bja/aew362. PMID 27940457
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Li J, Zhu H, Liao R. Enhanced recovery after surgery (ERAS) pathway for primary hip and knee arthroplasty: study protocol for a randomized controlled trial. Trials. 2019 Oct 22;20(1):599. doi: 10.1186/s13063-019-3706-8. PMID 31640757
- [Background] Kaye AD, Urman RD, Cornett EM, Hart BM, Chami A, Gayle JA, Fox CJ. Enhanced recovery pathways in orthopedic surgery. J Anaesthesiol Clin Pharmacol. 2019 Apr;35(Suppl 1):S35-S39. doi: 10.4103/joacp.JOACP_35_18. PMID 31142957
- [Background] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Background] Zhang XY, Ma JB. The efficacy of fascia iliaca compartment block for pain control after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Jan 25;14(1):33. doi: 10.1186/s13018-018-1053-1. PMID 30683117
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Sahoo RK, Jadon A, Sharma SK, Nair AS. Pericapsular nerve group (PENG) block for hip fractures: Another weapon in the armamentarium of anesthesiologists. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):295-296. doi: 10.4103/joacp.JOACP_295_20. Epub 2021 Jul 15. No abstract available. PMID 34349384
- [Background] Allard C, Pardo E, de la Jonquiere C, Wyniecki A, Soulier A, Faddoul A, Tsai ES, Bonnet F, Verdonk F. Comparison between femoral block and PENG block in femoral neck fractures: A cohort study. PLoS One. 2021 Jun 4;16(6):e0252716. doi: 10.1371/journal.pone.0252716. eCollection 2021. PMID 34086782
- [Background] Kukreja P, Avila A, Northern T, Dangle J, Kolli S, Kalagara H. A Retrospective Case Series of Pericapsular Nerve Group (PENG) Block for Primary Versus Revision Total Hip Arthroplasty Analgesia. Cureus. 2020 May 19;12(5):e8200. doi: 10.7759/cureus.8200. PMID 32572357
- [Background] Talawar P, Tandon S, Tripathy DK, Kaushal A. Combined pericapsular nerve group and lateral femoral cutaneous nerve blocks for surgical anaesthesia in hip arthroscopy. Indian J Anaesth. 2020 Jul;64(7):638-640. doi: 10.4103/ija.IJA_57_20. Epub 2020 Jul 1. No abstract available. PMID 32792743
- [Background] Thallaj A. Combined PENG and LFCN blocks for postoperative analgesia in hip surgery-A case report. Saudi J Anaesth. 2019 Oct-Dec;13(4):381-383. doi: 10.4103/sja.SJA_299_19. PMID 31572090
- [Background] 17. Kim YS, Park JM, Moon YS, Han SH. Assessment of pain in the elderly: A literature review. Natl Med J India. 2017;30(4):203-207. doi:10.4103/0970-258X.218673 El-Boghdadly K, Pawa A, Chin KJ. Local anesthetic systemic toxicity: current perspectives. Local Reg Anesth. 2018;11:35-44. Published 2018 Aug 8. doi:10.2147/LRA.S15451